CLINICAL TRIAL: NCT04223856
Title: An Open-label, Randomized, Controlled Phase 3 Study of Enfortumab Vedotin in Combination With Pembrolizumab Versus Chemotherapy Alone in Previously Untreated Locally Advanced or Metastatic Urothelial Cancer
Brief Title: Enfortumab Vedotin and Pembrolizumab vs. Chemotherapy Alone in Untreated Locally Advanced or Metastatic Urothelial Cancer
Acronym: EV-302
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry); Seagen Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGN22E-003; 2019-004542-15 (EudraCT Number); MK-3475-A39 (Other: Merck); KEYNOTE KN-A39 (Other: Merck); jRCT2031200284 (Registry Identifier: Japan Registry of Clinical Trials (jRCT)); CTR20220974 (Other: ChinaDrugTrials.org.cn)
Expanded Access: NCT04136808 (Approved for marketing)
Record Dates: First submitted 2020-01-06; First posted 2020-01-10 (Actual); Results first posted 2024-09-27 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Urothelial Cancer
Keywords: Urothelial Cancer; Enfortumab vedotin; metastatic urothelial cancer; pembrolizumab; locally advanced urothelial cancer
MeSH Terms: interventions — enfortumab vedotin; pembrolizumab; Cisplatin; Carboplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Enfortumab vedotin + pembrolizumab
  Interventions: Drug: Enfortumab vedotin; Drug: Pembrolizumab
- Arm B (Active Comparator): Gemcitabine + cisplatin or carboplatin
  Interventions: Drug: Cisplatin; Drug: Carboplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Enfortumab vedotin — Enfortumab vedotin administered as an IV infusion on Days 1 and 8 of every 3-week cycle
  Other Names: ASG-22CE; ASG-22ME; PADCEV
  Arms: Arm A
Drug: Pembrolizumab — IV infusion on Day 1 of every 3-week cycle
  Other Names: Keytruda
  Arms: Arm A
Drug: Cisplatin — administered as IV infusion on Day 1 of each 3-week cycle
  Arms: Arm B
Drug: Carboplatin — Dosed according to local guidelines and will be administered as IV infusion on Day 1 of each 3-week cycle
  Arms: Arm B
Drug: Gemcitabine — IV infusion on Days 1 and 8 of every 3 week cycle
  Arms: Arm B

SUMMARY:
This study is being done to see how well two drugs (enfortumab vedotin and pembrolizumab) work together to treat patients with urothelial cancer. The study will compare these drugs to other drugs that are usually used to treat this cancer (standard of care). The patients in this study will have cancer that has spread from their urinary system to other parts of their body.

DETAILED DESCRIPTION:
Japan PMDA has approved enfortumab vedotin (Padcev) for the treatment of advanced urothelial cancer. The study will continue as a post marketing study in Japan.

This study is being conducted to evaluate the combination of enfortumab vedotin + pembrolizumab versus standard of care gemcitabine + platinum-containing chemotherapy, in subjects with previously untreated locally advanced or metastatic urothelial cancer.

Enfortumab vedotin may be administered for an unlimited number of cycles until a protocol defined reason for study discontinuation occurs. Pembrolizumab may be administered for a maximum of 35 cycles or a protocol-defined reason for study discontinuation occurs, whichever is first. Cisplatin or carboplatin plus gemcitabine may be administered for a maximum of 6 cycles or a protocol-defined reason for study discontinuation occurs, whichever is first.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented, unresectable locally advanced or metastatic urothelial carcinoma
* Measurable disease by investigator assessment according to RECIST v1.1

  * Participants with prior definitive radiation therapy must have measurable disease per RECIST v1.1 that is outside the radiation field or has demonstrated unequivocal progression since completion of radiation therapy
* Participants must not have received prior systemic therapy for locally advanced or metastatic urothelial carcinoma with the following exceptions:

  * Participants that received neoadjuvant chemotherapy with recurrence >12 months from completion of therapy are permitted
  * Participants that received adjuvant chemotherapy following cystectomy with recurrence >12 months from completion of therapy are permitted
* Must be considered eligible to receive cisplatin- or carboplatin-containing chemotherapy, in the investigator's judgment
* Archival tumor tissue comprising muscle-invasive urothelial carcinoma or a biopsy of metastatic urothelial carcinoma must be provided for PD-L1 testing prior to randomization
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0, 1, or 2
* Adequate hematologic and organ function

Exclusion Criteria:

* Previously received enfortumab vedotin or other monomethyl auristatin E (MMAE)-based antibody-drug conjugate (ADCs)
* Received prior treatment with a programmed cell death ligand-1 (PD-(L)-1) inhibitor for any malignancy, including earlier stage urothelial cancer (UC), defined as a PD-1 inhibitor or PD-L1 inhibitor
* Received prior treatment with an agent directed to another stimulatory or co inhibitory T-cell receptor
* Received anti-cancer treatment with chemotherapy, biologics, or investigational agents not otherwise prohibited by exclusion criterion 1-3 that is not completed 4 weeks prior to first dose of study treatment
* Uncontrolled diabetes
* Estimated life expectancy of less than 12 weeks
* Active central nervous system (CNS) metastases
* Ongoing clinically significant toxicity associated with prior treatment that has not resolved to ≤ Grade 1 or returned to baseline
* Currently receiving systemic antimicrobial treatment for active infection (viral, bacterial, or fungal) at the time of randomization. Routine antimicrobial prophylaxis is permitted.
* Known active hepatitis B, active hepatitis C, or human immunodeficiency virus (HIV) infection.
* History of another invasive malignancy within 3 years before the first dose of study drug, or any evidence of residual disease from a previously diagnosed malignancy
* Documented history of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction, or cardiac symptoms consistent with New York Heart Association (NYHA) Class IV within 6 months prior to randomization
* Receipt of radiotherapy within 2 weeks prior to randomization
* Received major surgery (defined as requiring general anesthesia and >24 hour inpatient hospitalization) within 4 weeks prior to randomization
* Known severe (≥ Grade 3) hypersensitivity to any enfortumab vedotin excipient contained in the drug formulation of enfortumab vedotin
* Active keratitis or corneal ulcerations
* History of autoimmune disease that has required systemic treatment in the past 2 years
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Prior allogeneic stem cell or solid organ transplant
* Received a live attenuated vaccine within 30 days prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 886 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2028-03-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Zejing Wang, MD, PhD, Study Director — Seagen Inc.; John Lu, MD, Study Director — Seagen Inc.
Locations (260):
- United States (34):
  - Ironwood Cancer & Research Centers - Chandler, Chandler, Arizona
  - Arizona Oncology Associates PD - HOPE, Tucson, Arizona
  - Providence St Joseph Medical Center, Burbank, California
  - City of Hope National Medical Center, Duarte, California
  - University of California Los Angeles Medical Center, Los Angeles, California
  - University of California Irvine - Newport, Orange, California
  - Rocky Mountain Cancer Centers - Aurora, Aurora, Colorado
  - University of Colorado Hospital / University of Colorado, Aurora, Colorado
  - Cancer Centers of Colorado - Denver, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Eastern CT Hematology and Oncology Associates, Norwich, Connecticut
  - Lombardi Cancer Center / Georgetown University Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Winship Cancer Institute / Emory University School of Medicine, Atlanta, Georgia
  - Georgia Cancer Specialists / Northside Hospital Cancer Institute, Marietta, Georgia
  - Louisiana State University/ East Jefferson General Hospital, Metairie, Louisiana
  - Maine Health Cancer Care, Biddeford, Maine
  - Johns Hopkins Medical Center, Baltimore, Maryland
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - New Mexico Cancer Center, Albuquerque, New Mexico
  - New York University (NYU) Cancer Institute, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Vidant Medical Center, Greenville, North Carolina
  - The Cleveland Clinic, Cleveland, Ohio
  - Toledo Clinic Cancer Center, Toledo, Ohio
  - Hillman Cancer Center / University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Saint Francis Hospital / Bon Secours - South Carolina, Greenville, South Carolina
  - West Cancer Center & Research Institute, Germantown, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - UT Health East Texas Hope Cancer Center, Tyler, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Seattle Cancer Care Alliance / University of Washington, Seattle, Washington
- Argentina (9):
  - Site AR54008, Buenos Aire
  - Site AR54011, CABA
  - Site AR54005, Córdoba
  - Site AR54006, La Rioja
  - Site AR54004, Mendoza
  - Site AR54001, Rosario
  - Site AR54002, San Miguel
  - Site AR54012, San Miguel de Tucumán
  - Site AR54003, Viedma
- Australia (6):
  - Site AU61003, Box Hill
  - Site AUS61001, Douglas
  - Site AUS61004, Heidelberg
  - Site AUS61002, Macquarie Park
  - Site AUS61006, South Australia
  - Site AU61005, South Brisbane
- Belgium (5):
  - Site BE32003, Brussels
  - Site BE32002, Ghent
  - Site BE32001, Liège
  - Site BE32007, Lueven
  - Site BE32006, Roeselare
- Canada (11):
  - Site CA11004, Calgary, Alberta
  - Site CA11003, Edmonton, Alberta
  - Site CA11006, Vancouver, British Columbia
  - Site CA11002, Hamilton, Ontario
  - Site CA11009, London, Ontario
  - Site CA11011, Oshawa, Ontario
  - Site CA11012, Toronto, Ontario
  - Site CA11005, Toronto, Ontario
  - Site CA11010, Montreal, Quebec
  - Site CA11001, Montreal, Quebec
  - Site CA11008, Québec
- China (30):
  - Site CN86009, Beijing
  - Site CN86001, Beijing
  - Site CN86004, Beijing
  - Site CN86005, Beijing
  - Site CN86015, Bengbu
  - Site CN86003, Changchun
  - Site CN86006, Changsha
  - Site CN86016, Changsha
  - Site CN86010, Chengdu
  - Site CN86024, Chongqing
  - Site CN86007, Chongqing
  - Site CN86028, Fuzhou
  - Site CN86002, Guangzhou
  - Site CN86020, Gunagzhou
  - Site CN86018, Hangzhou
  - Site CN86013, Hangzhou
  - Site CN86022, Hangzhou
  - Site CN86025, Hefei
  - Site CN86027, Jinan
  - Site CN86017, Nanjing
  - Site CN86012, Nanjing
  - Site CN86021, Ningbo
  - Site CN86014, Shanghai
  - Site CN86011, Shenyang
  - Site CN86023, Tianjin
  - Site CN86019, Tianjin
  - Site CN86029, Wenzhou
  - Site CN86008, Wuhan
  - Site CN86030, Xicheng District
  - Site CN86026, Xuzhou
- Czechia (4):
  - Site CZ42006, Brno
  - Site CZ42001, Hradec Králové
  - Site CZ42004, Olomouc
  - Site CZ42005, Praha 4-Krc
- Denmark (2):
  - Site DK45001, Aalborg
  - Site DK45003, Aarhus N
- France (7):
  - Site FR33014, Bordeaux
  - Site FR33016, Lyon
  - Site FR33003, Nice
  - Site FR33020, Pierre-Bénite
  - Site FR33013, Strasbourg
  - Site FR33017, Tours
  - Site FR33011, Villejuif-Cedex-France
- Germany (16):
  - Site DE49003, Berlin
  - Site DE49013, Bielefeld
  - Site DE49016, Düsseldorf
  - Site DE49014, Erlangen
  - Site DE49011, Essen
  - Site DE49007, Frankfurt am Main
  - Site DE49015, Göttingen
  - Site DE49005, Heidelberg
  - Site DE49009, Herne
  - Site DE49006, Jena
  - Site DE49001, Lübeck
  - Site DE49008, Magdeburg
  - Site DE49012, Mannheim
  - Site DE49002, München
  - Site DE49004, Tübingen
  - Site DE49010, Ulm
- Hungary (5):
  - Site HU36003, Budapest
  - Site HU36002, Budapest
  - Site HU36006, Debrecen
  - Site HU36001, Nyíregyháza
  - Site HU36005, Szolnok
- Israel (10):
  - Site IL97203, Beersheba
  - Site IL97201, Haifa
  - Site IL97209, Holon
  - Site IL97206, Jerusalem
  - Site IL97202, Kfar Saba
  - Site IL97208, Petah Tikva
  - Site IL97211, Rehovot
  - Site IL97210, Tel Aviv
  - Site IL97204, Tel Litwinsky
  - Site IL97205, Ẕerifin
- Italy (11):
  - Site IT39005, Areezo
  - Site IT39008, Candiolo
  - Site IT39009, Cremona
  - Site IT39006, Genova
  - Site IT39003, Meldola
  - Site IT39014, Milan
  - Site IT39007, Milan
  - Site IT39004, Pisa
  - Site IT39002, Terni
  - Site IT39011, Torrette
  - Site IT39001, Verona
- Japan (20):
  - Site JP81002, Bunkyō City
  - Site JP81009, Chiba
  - Site JP81018, Chiba
  - Site JP81013, Fukuoka
  - Site JP81020, Fukuoka
  - Site JP81011, Hirosaki
  - Site JP81006, Kawasaki-shi
  - Site JP81001, Kōtoku
  - Site JP81017, Kyoto
  - Site JP81015, Niigata
  - Site JP81005, Okayama
  - Site JP81008, Osaka
  - Site JP81016, Osakasayama-Shi
  - Site JP81007, Sapporo
  - Site JP81012, Sendai
  - Site JP81014, Tokushima
  - Site JP81019, Tokyo
  - Site JP81003, Toyama
  - Site JP81004, Tsukuba
  - Site JP81010, Ube
- Netherlands (7):
  - Site NL31002, Amsterdam
  - Site NL31001, Amsterdam
  - Site NL31005, Amsterdam, Noord-Holland
  - Site NL31007, Leeuwarden
  - Site NL31004, Nieuwegein
  - Site NL31003, Rotterdam
  - Site NL31006, Utrecht
- Site PL48002, Warsaw, Poland
- Russia (18):
  - Site RU70016, Arkhangelsk
  - Site RU70013, Barnaul
  - Site RU70020, Ivanovo
  - Site RU70014, Krasnoyarsk
  - Site RU70006, Leningradskaya Oblast'
  - Site RU70004, Moscow
  - Site RU70011, Moscow
  - Site RU70003, Moscow
  - Site RU70017, Nizhny Novgorod
  - Site RU70002, Omsk
  - Site RU70019, Pyatigorsk
  - Site RU70010, Saint Petersburg
  - Site RU70007, Saint Petersburg
  - Site RU70008, Saint Petersburg
  - Site RU70012, Saint Petersburg
  - Site RU70009, Saransk
  - Site RU70015, Tyumen
  - Site RU70005, Ufa
- Singapore (3):
  - Site SG65001, Singapore
  - Site SG65002, Singapore
  - Site SG65003, Singapore
- South Korea (8):
  - Site KR82001, Daejeon
  - Site KR82002, Goyang-si
  - Site KR82008, Hwasun
  - Site KR82004, Seongnam-si
  - Site KR82003, Seoul
  - Site KR82005, Seoul
  - Site KR82007, Seoul
  - Site KR82006, Seoul
- Spain (18):
  - Site ES34017, Barcelona
  - Site ES34010, Barcelona
  - Site ES34006, Barcelona
  - Site ES34001, Barcelona
  - Site ES34008, Barcelona
  - Site ES34013, Córdoba
  - Site ES34021, Lugo
  - Site ES34018, Madrid
  - Site ES34002, Madrid
  - Site ES34003, Madrid
  - Site ES34015, Madrid
  - Site ES34004, Manresa
  - Site ES34020, Pamplona
  - Site ES34016, Sabadell
  - Site ES34012, Santander
  - Site ES34007, Seville
  - Site ES34019, Valencia
  - Site ES34009, Valencia
- Switzerland (4):
  - Site CH41004, Basel
  - Site CH41002, Bern
  - Site CH41001, Chur
  - Site CH41003, Winterthur
- Taiwan (7):
  - Site TW88603, Kaohsiung City
  - Site TW88602, Kweishan
  - Site TW88607, Taichung
  - Site TW88606, Taichung
  - Site TW88604, Tainan
  - Site TW88605, Taipei
  - Site TW88601, Taipei
- Thailand (7):
  - Site TH66004, Bangkok
  - Site TH66003, Bangkok
  - Site TH66006, Bangkok
  - Site TH66005, Chiang Mai
  - Site TH66002, Hat Yai
  - Site TH66007, Muang
  - Site TH66001, Ratchathewi
- Turkey (Türkiye) (9):
  - Site TR90007, Ankara
  - Site TR90009, Ankara
  - Site TR90005, Antalya
  - Site TR90004, Edirne
  - Site TR90008, Istanbul
  - Site TR90003, Istanbul
  - Site TR90002, Istanbul
  - Site TR90001, Konya
  - Site TR90006, Malatya
- United Kingdom (8):
  - Site UK44005, Glasgow
  - Site UK44001, London
  - Site UK44009, London
  - Site UK44006, Oxford
  - Site UK44010, Plymouth
  - Site UK44002, Preston
  - Site UK44003, Sheffield
  - Site UK44008, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kikuchi E, Van der Heijden MS, Valderrama BP, Gupta S, Bedke J, Shin SJ, Li JR, Guo J, Danchaivijitr P, Kanesvaran R, Park SH, Su WP, Kandori S, Bae WK, Wong A, Gorla S, Bavle A, Yu X, Lu YT, Powles T. Pan-Asian subgroup analysis of EV-302/KEYNOTE-A39: a phase 3 study to evaluate enfortumab vedotin and pembrolizumab in patients with untreated advanced urothelial carcinoma. Int J Clin Oncol. 2026 Jan 21. doi: 10.1007/s10147-025-02950-8. Online ahead of print. PMID 41563650
- [Derived] Meng Y, Zhang S, Aout M, Babcock A, Li H, Lai Y, Brand-Wiita S, Notinger S, Bavle A, Mamtani R. Cost-effectiveness of enfortumab vedotin plus pembrolizumab as a first-line treatment of locally advanced or metastatic urothelial carcinoma in the United States. J Med Econ. 2025 Dec;28(1):1779-1797. doi: 10.1080/13696998.2025.2567190. Epub 2025 Oct 14. PMID 41039930
- [Derived] Gupta S, Loriot Y, Van der Heijden MS, Bedke J, Valderrama BP, Kikuchi E, Flechon A, Petrylak D, De Santis M, Galsky MD, Lee JL, Swami U, Sridhar SS, De Giorgi U, Wright P, Shih V, Lu YT, Guan X, Dillon R, Shetty A, Moreno BH, Beaumont JL, Purnajo I, McManus S, Powles T. Enfortumab vedotin plus pembrolizumab versus chemotherapy in patients with previously untreated locally advanced or metastatic urothelial cancer (EV-302): patient-reported outcomes from an open-label, randomised, controlled, phase 3 study. Lancet Oncol. 2025 Jun;26(6):795-805. doi: 10.1016/S1470-2045(25)00158-5. PMID 40449498
- [Derived] Niegisch G. Enfortumab Vedotin and Pembrolizumab - A New Perspective on Urothelial Cancer. N Engl J Med. 2024 Mar 7;390(10):944-946. doi: 10.1056/NEJMe2400311. No abstract available. PMID 38446680
- [Derived] Powles T, Valderrama BP, Gupta S, Bedke J, Kikuchi E, Hoffman-Censits J, Iyer G, Vulsteke C, Park SH, Shin SJ, Castellano D, Fornarini G, Li JR, Gumus M, Mar N, Loriot Y, Flechon A, Duran I, Drakaki A, Narayanan S, Yu X, Gorla S, Homet Moreno B, van der Heijden MS; EV-302 Trial Investigators. Enfortumab Vedotin and Pembrolizumab in Untreated Advanced Urothelial Cancer. N Engl J Med. 2024 Mar 7;390(10):875-888. doi: 10.1056/NEJMoa2312117. PMID 38446675
- [Derived] Hoimes CJ, Flaig TW, Milowsky MI, Friedlander TW, Bilen MA, Gupta S, Srinivas S, Merchan JR, McKay RR, Petrylak DP, Sasse C, Moreno BH, Yu Y, Carret AS, Rosenberg JE. Enfortumab Vedotin Plus Pembrolizumab in Previously Untreated Advanced Urothelial Cancer. J Clin Oncol. 2023 Jan 1;41(1):22-31. doi: 10.1200/JCO.22.01643. Epub 2022 Aug 30. PMID 36041086

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with untreated locally advanced or metastatic urothelial cancer (UC) were enrolled in the study.
Pre-assignment Details: Results are reported only for primary outcome measures at primary completion date (08-Aug-2023). Remaining secondary outcome measures whose analysis are not final, results would be reported at study completion date.
Groups:
- Enfortumab Vedotin + Pembrolizumab: Participants received enfortumab vedotin at 1.25 milligram per kilogram (mg/kg) as an intravenous (IV) infusion over approximately 30 minutes on Days 1 and 8 of each cycle, and pembrolizumab 200 mg as an IV infusion over approximately 30 minutes on Day 1 of each cycle, after completion of the enfortumab vedotin infusion. 1 cycle = 3 weeks.
- Standard of Care: Participants received gemcitabine at 1000 mg/m^2 as an IV infusion on Days 1 and 8 of each cycle, and either cisplatin (70 mg/m^2) or carboplatin (area under curve [AUC] 4.5, or AUC 5 according to local guidelines) on Day 1 of each cycle, with adequate pre- and post-hydration, by IV infusion per institutional standards. 1 cycle = 3 weeks.
Period: Overall Study
Arm/Group | Enfortumab Vedotin + Pembrolizumab | Standard of Care
Started | 442 | 444
Treated | 440 | 433
Completed | 8 | 244
Not Completed | 434 | 200
Not completed — Progressive disease | 153 | 73
Not completed — Adverse Event | 97 | 62
Not completed — Physician Decision | 9 | 28
Not completed — Withdrawal by Subject | 22 | 24
Not completed — Other | 7 | 2
Not completed — Randomized but not treated | 2 | 11
Not completed — On-treatment | 144 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) analysis set include all randomized participants. Participants were analyzed according to the treatment arm assigned at randomization regardless of the actual treatment received.
Groups:
- Enfortumab Vedotin + Pembrolizumab: Participants received enfortumab vedotin at 1.25 mg/kg as an IV infusion over approximately 30 minutes on Days 1 and 8 of each cycle, and pembrolizumab 200 mg as an IV infusion over approximately 30 minutes on Day 1 of each cycle, after completion of the enfortumab vedotin infusion. 1 cycle = 3 weeks.
- Standard of Care: Participants received gemcitabine at 1000 mg/m^2 as an IV infusion on Days 1 and 8 of each cycle, and either cisplatin (70 mg/m^2) or carboplatin (AUC 4.5, or AUC 5 according to local guidelines) on Day 1 of each cycle, with adequate pre- and post-hydration, by IV infusion per institutional standards. 1 cycle = 3 weeks.
- Total: Total of all reporting groups
Arm/Group | Enfortumab Vedotin + Pembrolizumab | Standard of Care | Total
Number analyzed (Participants) | 442 | 444 | 886
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.9 (9.1) | 68.0 (9.4) | 67.9 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 108 | 206
  Male | 344 | 336 | 680
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 52 | 52 | 104
  Not Hispanic or Latino | 359 | 343 | 702
  Unknown or Not Reported | 31 | 49 | 80
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 2 | 2 | 4
  Race: Asian | 99 | 92 | 191
  Race: Black or African American | 3 | 7 | 10
  Race: Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Race: White | 308 | 290 | 598
  Race: Other | 3 | 1 | 4
  Race: Multiple | 0 | 4 | 4
  Race: Unknown | 5 | 10 | 15
  Race: Not Reported | 22 | 37 | 59

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors (RECIST) Version (v) 1.1 by Blinded Independent Central Review (BICR)
Description: PFS was defined as the time from date of randomization to first documentation of disease progression (PD), or to death due to any cause, whichever occurred first. PD: at least a 20 percent (%) increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeter (mm). PD could also be unequivocal progression of non-target lesions or the presence of unequivocal new lesions. Kaplan-Meier method was used for analysis.
Time Frame: From the date of randomization to first documentation of PD or death due to any cause, whichever occurred first (maximum exposure to treatment was up to 39.2 months)
Population: ITT analysis set included all randomized participants. Participants were analyzed according to the treatment arm assigned at randomization regardless of the actual treatment received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enfortumab Vedotin + Pembrolizumab | Standard of Care
Number analyzed (Participants) | 442 | 444
Months | 12.5 [10.4 to 16.6] | 6.3 [6.2 to 6.5]
Statistical Analysis 1: Comparison: Enfortumab Vedotin + Pembrolizumab vs Standard of Care; Test type: Superiority; p < 0.00001, Log Rank — P value was calculated using stratified log-rank test. The p-value threshold for statistical significance is 0.005; Hazard Ratio (HR) = 0.450, 95% CI 2-sided [0.377 to 0.538] — HR was calculated using stratified Cox proportional hazards model

2. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death from any cause. In the absence of death, OS was censored at the date the participant was last known to be alive. Kaplan-Meier method was used for analysis.
Time Frame: From randomization to date of death due to any cause or censoring date, whichever occurred first (maximum exposure to treatment was up to 39.2 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enfortumab Vedotin + Pembrolizumab | Standard of Care
Number analyzed (Participants) | 442 | 444
Months | 31.5 [25.4 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with event. | 16.1 [13.9 to 18.3]
Statistical Analysis 1: Comparison: Enfortumab Vedotin + Pembrolizumab vs Standard of Care; Test type: Superiority — P value was calculated using stratified log-rank test. The p-value threshold for statistical significance is 0.01548; p < 0.00001, Log Rank; Hazard Ratio (HR) = 0.468, 95% CI 2-sided [0.376 to 0.582] — HR was calculated using stratified Cox proportional hazards model

3. Secondary Outcome: Percentage of Participants With Objective Response Rate (ORR) Per RECIST v1.1 by BICR
Description: ORR as per RECIST v1.1 by BICR was defined as the percentage of participants with confirmed complete response (CR) or partial response (PR) CR was defined as disappearance of all lesions including non-target lesions (not just target lesions). Any pathological lymph nodes must have reduction in short axis to<10 mm. PR was defined as at least 30 percent [%] decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. For a response to be considered as confirmed, the subsequent response needs to be at least 4 weeks after the initial response.
Time Frame: From first dose till CR/PR or PD or death, whichever occurred first (maximum up to approximately 7.4 years)
Reporting Status: Not Posted, anticipated posting 2027-09

4. Secondary Outcome: Time to Pain Progression (TTPP)
Description: TTPP was defined as the time from the date of randomization to date of pain progression. Pain progression was defined as a participant reporting either of the following, whichever came first: 1) Increase of 2 or more points from baseline on Brief Pain Inventory - Short Form (BPI-SF) Question 3 (i.e., pain at its worst in the last 24 hours, score range 0 to 10 with higher scores associated with higher pain levels) maintained for at least two consecutive assessments. 2) Initiation of new opioid medication from baseline for pain with usage maintained for at least two consecutive assessments as recorded in BPI-SF Question 7 (i.e., What medications received for pain).
Time Frame: From the date of randomization to date of pain progression (maximum up to approximately 7.4 years)
Reporting Status: Not Posted, anticipated posting 2027-09

5. Secondary Outcome: Change From Baseline in Worst Pain Using BPI-SF at Week 26
Description: Brief Pain Inventory (BPI-SF) was defined as summary of the worst, least, and average pain experienced in the last 24 hours as well as pain right now and number of pain locations were provided for each treatment arm. BPI-sf worst pain measured the severity of pain based on the pain at its worst in the last 24 hours, score range 0 to 10 with higher scores associated with higher pain levels.
Time Frame: Baseline, Week 26
Reporting Status: Not Posted, anticipated posting 2027-09

6. Secondary Outcome: PFS Per RECIST v1.1 by Investigator Assessment
Description: PFS as per RECIST v1.1 by investigator was defined as the time from date of randomization to first documentation of PD, or to death due to any cause, whichever comes first. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. PD could also be unequivocal progression of non-target lesions or the presence of unequivocal new lesions.
Time Frame: From the date of randomization to first documentation of PD or death due to any cause, whichever occurred first (maximum up to approximately 7.4 years)
Reporting Status: Not Posted, anticipated posting 2027-09

7. Secondary Outcome: ORR Per RECIST v1.1 by Investigator Assessment
Description: ORR as per RECIST v1.1 by investigator was defined as the percentage of participants with confirmed CR or PR. CR was defined as disappearance of all lesions including non-target lesions (not just target lesions). Any pathological lymph nodes must have reduction in short axis to<10 mm. PR was defined as at least 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. For a response to be considered as confirmed, the subsequent response needs to be at least 4 weeks after the initial response.
Time Frame: From first dose till CR/PR or PD or death, whichever occurred first (maximum up to approximately 7.4 years)
Reporting Status: Not Posted, anticipated posting 2027-09

8. Secondary Outcome: Duration of Response (DOR) Per RECIST v1.1 by BICR
Description: DOR was defined as the time from the first objective response (CR or PR that is subsequently confirmed) to the first documented PD per RECIST v1.1 per BICR or death from any cause, whichever occurs first. DOR will only include subjects with a confirmed response (CR or PR per RECIST v1.1). CR was defined as disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to<10 mm. PR was defined as at least 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. For a response to be considered as confirmed, the subsequent response needs to be at least 4 weeks after the initial response. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From the date of first documented response of CR or PR to the first documented disease progression or to death from any cause, whichever occurred first (maximum up to approximately 7.4 years)
Reporting Status: Not Posted, anticipated posting 2027-09

9. Secondary Outcome: DOR Per RECIST v1.1 by Investigator Assessment
Description: DOR was defined as the time from the first objective response (CR or PR that is subsequently confirmed) to the first documented PD per RECIST v1.1 per investigator or death from any cause, whichever occurs first. DOR will only include subjects with a confirmed response (CR or PR per RECIST v1.1). CR was defined as disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to<10 mm. PR was defined as at least 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. For a response to be considered as confirmed, the subsequent response needs to be at least 4 weeks after the initial response.
Time Frame: as for outcome 8
Reporting Status: Not Posted, anticipated posting 2027-09

10. Secondary Outcome: Disease Control Rate (DCR) Per RECIST v1.1 by BICR
Description: DCR by BICR was defined as the percentage of participants with confirmed response (CR or PR), or SD (or non-CR/non-PD), per RECIST v1.1. Subjects who have no post-baseline response assessments will be considered as non-responders for calculating the DCR. Only response assessments before the first documented PD or subsequent anticancer therapies were considered. CR was defined as disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to<10 mm. PR was defined as at least 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. For a response to be considered as confirmed, the subsequent response needs to be at least 4 weeks after the initial response. SD was defined as a change in tumor size that is neither radiological response (>30% shrinkage) nor progression (>20% growth).
Time Frame: From the date of randomization to the date of PD or death from any cause or censoring date, whichever occurred first (maximum up to approximately 7.4 years)
Reporting Status: Not Posted, anticipated posting 2027-09

11. Secondary Outcome: DCR Per RECIST v1.1 by Investigator Assessment
Description: as for outcome 10
Time Frame: as for outcome 10
Reporting Status: Not Posted, anticipated posting 2027-09

12. Secondary Outcome: Mean Scores in Patient Reported Outcome (PRO) Assessment Measured by the EuroQOL Five Dimensions Questionnaire 5L (EQ-5D-5L)
Description: The EQ-5D-5L is a 5-item self-reported measure of functioning and well-being, which assesses 5 dimensions of health, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression (EQ-5D-5L User Guide, 2019). Each dimension comprises 5 levels (no problems, slight problems, moderate problems, severe problems, and extreme problems).
Time Frame: End of study (approximately up to 7.4 years)
Reporting Status: Not Posted, anticipated posting 2027-09

13. Secondary Outcome: Change From Baseline in PRO Assessment Measured by the EQ-5D-5L
Description: as for outcome 12
Time Frame: Baseline, End of study (approximately up to 7.4 years)
Reporting Status: Not Posted, anticipated posting 2027-09

14. Secondary Outcome: Mean Scores in PRO Assessment Measured by European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30)
Description: EORTC QLQ-C30: included functional scales (physical, role, cognitive, emotional, and social), global health status (GHS), symptom scales (fatigue, pain, nausea/vomiting), and single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea, and financial difficulties). Most questions used 4- point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores averaged, transformed to 0- 100 scale; higher score=better level of functioning or greater degree of symptoms.
Time Frame: End of study (approximately up to 7.4 years)
Reporting Status: Not Posted, anticipated posting 2027-09

15. Secondary Outcome: Change From Baseline in PRO Assessment Measured by EORTC QLQ-C30
Description: EORTC QLQ-C30: included functional scales (physical, role, cognitive, emotional, and social), global health status (GHS), symptom scales (fatigue, pain, nausea/vomiting), and single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea, and financial difficulties). Most questions used 4- point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores averaged, transformed to 0- 100 scale; higher score=better level of functioning or greater degree of symptoms. Change from baseline=Cycle/Day score minus baseline score.
Time Frame: Baseline, End of study (approximately up to 7.4 years)
Reporting Status: Not Posted, anticipated posting 2027-09

16. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent are events between first dose of study drug and up to 37 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From start of treatment up to 37 days after last dose of study drug (approximately up to 7.4 years)
Reporting Status: Not Posted, anticipated posting 2027-09

17. Secondary Outcome: Number of Participants With Serious TEAE
Description: SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/ incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 37 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From start of treatment up to 37 days after last dose of study drug (approximately up to 7.4 years)
Reporting Status: Not Posted, anticipated posting 2027-09

18. Secondary Outcome: Number of Participants With Grade 3-5 TEAE
Description: AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. As per common terminology criteria for adverse events (CTCAE) version 4, Grade 3= severe AE; Grade 4= life-threatening or disabling AE; Grade 5= death related to an AE.
Time Frame: From start of treatment up to 37 days after last dose of study drug (approximately up to 7.4 years)
Reporting Status: Not Posted, anticipated posting 2027-09

19. Secondary Outcome: Number of Participants Related to Treatment AEs
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment relatedness was assessed by the investigator.
Time Frame: From start of treatment up to 37 days after last dose of study drug (approximately up to 7.4 years)
Reporting Status: Not Posted, anticipated posting 2027-09

20. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Laboratory abnormalities included Hematology and Serum Chemistry. In Hematology (increased : hemoglobin, lymphocytes, leukocytes, and decreased : hemoglobin, lymphocytes, neutrophils, platelets and leukocytes) and In serum chemistry (increased in : alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, bilirubin, calcium corrected for albumin, creatinine, glucose (non-fasting), potassium, sodium, and decreased in albumin, calcium corrected for albumin, glucose (non-fasting), potassium, phosphate and sodium).
Time Frame: From start of treatment up to 37 days after last dose of study drug (approximately up to 7.4 years)
Reporting Status: Not Posted, anticipated posting 2027-09

21. Secondary Outcome: Number of Participants With Treatment Discontinuation Rate Due to AEs
Time Frame: During study (approximately up to 7.4 years)
Reporting Status: Not Posted, anticipated posting 2027-09

ADVERSE EVENTS:
Time Frame: From start of treatment up to 37 days after last dose of study drug (up to 40 months 9 days)
Description: Same event may appear as both non-serious adverse event (SAE) and SAE; however, what is presented are distinct events. An event may be categorized as serious in 1 participant and non-serious in other participant, or a participant may have experienced both SAE and non-SAE. Data for all-cause mortality was collected for all enrolled participants, data for SAE and non-SAE were collected for treated participants.
Arm/Group | Enfortumab Vedotin + Pembrolizumab | Standard of Care
All-Cause Mortality (participants affected / at risk) | 133/442 | 226/444
Serious Adverse Events (participants affected / at risk) | 220/440 | 169/433
Other Adverse Events (participants affected / at risk) | 435/440 | 418/433
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enfortumab Vedotin + Pembrolizumab (N=440) | Standard of Care (N=433)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 17 (18)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 12 (12)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 7 (7)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 13 (13)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2)
Acute right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 4 (4)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure (Cardiac disorders) | 3 (3) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Immune-mediated myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Myocarditis (Cardiac disorders) | 2 (3) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 2 (2) | 0 (0)
Hypercalcaemia of malignancy (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 8 (8) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 3 (4) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 14 (15) | 2 (2)
Duodenal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 2 (2) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1)
Large intestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Malignant gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (5) | 4 (4)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (7) | 2 (2)
Asthenia (General disorders) | 3 (3) | 4 (5)
Condition aggravated (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 3 (3)
General physical health deterioration (General disorders) | 1 (1) | 7 (8)
Malaise (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Performance status decreased (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 9 (10) | 10 (15)
Sudden death (General disorders) | 1 (1) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis sclerosing (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 3 (3) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 3 (3) | 0 (0)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 8 (8) | 5 (5)
COVID-19 pneumonia (Infections and infestations) | 5 (5) | 3 (3)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus colitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 3 (3) | 2 (2)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 2 (2) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (2)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 2 (2)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Pelvic infection (Infections and infestations) | 1 (1) | 0 (0)
Perineal abscess (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 10 (10) | 5 (5)
Pneumonia aspiration (Infections and infestations) | 3 (3) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 4 (4) | 6 (6)
Pyelonephritis acute (Infections and infestations) | 1 (4) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Sepsis (Infections and infestations) | 7 (7) | 8 (8)
Septic shock (Infections and infestations) | 3 (3) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 16 (16) | 31 (39)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 2 (2) | 5 (5)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Alanine aminotransferase increased (Investigations) | 5 (5) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 2 (2)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 4 (4)
Prothrombin time prolonged (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (4) | 5 (5)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercreatininaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (6) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (6) | 5 (6)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1)
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic hyperglycaemic coma (Nervous system disorders) | 1 (1) | 0 (0)
Immune-mediated encephalitis (Nervous system disorders) | 1 (1) | 0 (0)
Immune-mediated neuropathy (Nervous system disorders) | 1 (2) | 0 (0)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0)
Optic neuritis (Nervous system disorders) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 23 (27) | 11 (13)
Calculus bladder (Renal and urinary disorders) | 2 (2) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 7 (7) | 10 (10)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 2 (2)
Immune-mediated nephritis (Renal and urinary disorders) | 2 (2) | 0 (0)
Postrenal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2) | 3 (3)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinoma (Renal and urinary disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal dyskinesia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (7)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute generalised exanthematous pustulosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 (7) | 0 (0)
Rash morbilliform (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
SJS-TEN overlap (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Toxic erythema of chemotherapy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 4 (4)
Hypotension (Vascular disorders) | 2 (2) | 1 (1)
Iliac artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Lymphocele (Vascular disorders) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enfortumab Vedotin + Pembrolizumab (N=440) | Standard of Care (N=433)
Anaemia (Blood and lymphatic system disorders) | 106 (168) | 255 (362)
Leukopenia (Blood and lymphatic system disorders) | 16 (25) | 47 (91)
Neutropenia (Blood and lymphatic system disorders) | 43 (70) | 178 (360)
Thrombocytopenia (Blood and lymphatic system disorders) | 19 (21) | 147 (266)
Tinnitus (Ear and labyrinth disorders) | 6 (6) | 29 (31)
Hypothyroidism (Endocrine disorders) | 45 (47) | 3 (3)
Cataract (Eye disorders) | 22 (23) | 1 (1)
Dry eye (Eye disorders) | 50 (52) | 5 (5)
Lacrimation increased (Eye disorders) | 36 (42) | 2 (2)
Vision blurred (Eye disorders) | 26 (28) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 44 (52) | 25 (30)
Constipation (Gastrointestinal disorders) | 116 (136) | 146 (168)
Diarrhoea (Gastrointestinal disorders) | 161 (237) | 67 (78)
Dry mouth (Gastrointestinal disorders) | 41 (41) | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 25 (26) | 18 (20)
Nausea (Gastrointestinal disorders) | 114 (144) | 176 (233)
Stomatitis (Gastrointestinal disorders) | 39 (46) | 27 (31)
Vomiting (Gastrointestinal disorders) | 48 (57) | 67 (95)
Asthenia (General disorders) | 75 (123) | 84 (112)
Fatigue (General disorders) | 152 (182) | 167 (199)
Oedema peripheral (General disorders) | 60 (72) | 47 (57)
Pyrexia (General disorders) | 72 (97) | 60 (72)
COVID-19 (Infections and infestations) | 55 (59) | 16 (16)
Conjunctivitis (Infections and infestations) | 27 (30) | 0 (0)
Urinary tract infection (Infections and infestations) | 76 (96) | 64 (92)
Alanine aminotransferase increased (Investigations) | 74 (123) | 33 (52)
Aspartate aminotransferase increased (Investigations) | 66 (106) | 27 (45)
Blood alkaline phosphatase increased (Investigations) | 22 (33) | 16 (19)
Blood creatinine increased (Investigations) | 37 (49) | 49 (58)
Neutrophil count decreased (Investigations) | 15 (20) | 56 (109)
Platelet count decreased (Investigations) | 4 (7) | 61 (94)
Weight decreased (Investigations) | 144 (152) | 38 (38)
White blood cell count decreased (Investigations) | 5 (8) | 25 (45)
Decreased appetite (Metabolism and nutrition disorders) | 142 (168) | 112 (136)
Hyperglycaemia (Metabolism and nutrition disorders) | 68 (101) | 11 (13)
Hypokalaemia (Metabolism and nutrition disorders) | 35 (57) | 25 (30)
Hypomagnesaemia (Metabolism and nutrition disorders) | 18 (27) | 27 (31)
Hyponatraemia (Metabolism and nutrition disorders) | 36 (54) | 26 (38)
Hypophosphataemia (Metabolism and nutrition disorders) | 30 (41) | 17 (20)
Arthralgia (Musculoskeletal and connective tissue disorders) | 57 (72) | 21 (23)
Back pain (Musculoskeletal and connective tissue disorders) | 50 (60) | 33 (33)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 28 (28) | 7 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 26 (30) | 11 (15)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 31 (37) | 23 (26)
Dizziness (Nervous system disorders) | 36 (38) | 43 (46)
Dysgeusia (Nervous system disorders) | 93 (106) | 37 (38)
Headache (Nervous system disorders) | 33 (42) | 26 (27)
Paraesthesia (Nervous system disorders) | 36 (39) | 8 (9)
Peripheral sensory neuropathy (Nervous system disorders) | 228 (271) | 44 (44)
Insomnia (Psychiatric disorders) | 45 (47) | 24 (24)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 23 (29)
Haematuria (Renal and urinary disorders) | 52 (67) | 34 (42)
Cough (Respiratory, thoracic and mediastinal disorders) | 54 (60) | 22 (23)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 22 (25) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 54 (63) | 47 (55)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 27 (27)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 29 (31)
Alopecia (Skin and subcutaneous tissue disorders) | 152 (154) | 34 (34)
Dry skin (Skin and subcutaneous tissue disorders) | 76 (84) | 6 (6)
Eczema (Skin and subcutaneous tissue disorders) | 28 (33) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 182 (259) | 29 (33)
Rash macular (Skin and subcutaneous tissue disorders) | 43 (57) | 6 (7)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 143 (208) | 15 (15)
Rash papular (Skin and subcutaneous tissue disorders) | 34 (42) | 3 (3)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 24 (27) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-09-29): https://cdn.clinicaltrials.gov/large-docs/56/NCT04223856/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-22): https://cdn.clinicaltrials.gov/large-docs/56/NCT04223856/SAP_001.pdf